CLINICAL TRIAL: NCT01731028
Title: Non-interventional, Observational Study of the Application of Zomacton® in the Treatment of Growth Hormone Deficiency in Routine Clinical Practice
Brief Title: Surveillance of Treatment of Children With Growth Hormone Deficiency With Zomacton®
Status: Withdrawn | Type: Observational
Why Stopped: Change of local requirements
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000091
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Somatropin: Children with growth hormone deficiency treated with somatropin as Zomacton® according to the marketing authorization
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Somatropin powder and solvent for solution for injection

SUMMARY:
The purpose of this study is to investigate the long-term treatment with Zomacton® for pituitary short stature in children with insufficient growth hormone production and/or short stature caused by Turner's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* therapeutic need according to the approved specific products characteristics (SPC)

Exclusion Criteria:

* contraindication according to the SPC

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with inadequate secretion of growth-hormone; growth retardation due to Turner's syndrome
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Zomacton® treatment measured by the increase in body height per annuum | 5 years

SECONDARY OUTCOMES:
Efficacy of Zomacton® treatment measured by the increase in body weight per annuum | 5 years
Safety of Zomacton® and the application device measured by local adverse reactions to the application device | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals